CLINICAL TRIAL: NCT04934202
Title: Cohort Follow-up at 6-12 Months of Survivors of Hospitalization for COVID-19 During the 2nd Wave of the Epidemic From a University Hospital in France
Brief Title: Cohort Follow-up of Survivors of Hospitalization for COVID-19 During the 2nd Wave of the Epidemic in France
Acronym: COMEBAC 2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: COMEBAC 2
Record Dates: First submitted 2021-06-18; First posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Sequelae; Fibrosis; Post-COVID Syndrome; Post-traumatic Stress Disorder
MeSH Terms: conditions — Fibrosis; Stress Disorders, Post-Traumatic | interventions — Remote Consultation; Ambulatory Care Facilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients from the 1st epidemic wave: One year after their discharge from the initial hospitalization, patients who presented symptoms during the evaluation in COMEBAC "1st wave" in summer 2020 will benefit from a telephone assessment on the same schedule as that detailed above. If symptoms persist, they will be called to the day hospital for an assessment similar to the one detailed above.
  Interventions: Other: Teleconsultation; Other: Outpatient clinic
- Patients from the 2nd epidemic wave: As during the evaluation carried out during the 1st wave, the detection of persistent symptoms will be done in two stages:
  * During a teleconsultation, to which all eligible patients will be invited, systematically looking for general, neurological, cognitive and respiratory symptoms
  * During a hospitalization in an outpatient clinic to which all survivors who have stayed in an intensive care unit (ICU) will be invited and, among patients who have not stayed in an ICU, those who have residual symptoms detected during the teleconsultation.
  Interventions: Other: Teleconsultation; Other: Outpatient clinic

INTERVENTIONS:
Other: Teleconsultation — Teleconsulting physicians will subject patients to a standardized questionnaire that will look for the following symptoms:
  * General signs: Anorexia, fatigue, new hospitalization, weight loss,
  * Respiratory signs: recent dyspnoea, chest discomfort, chest pain, new cough, abnormal lung CT scan since discharge
  * Neurological signs: headache, paraesthesia, anosmia, limb paralysis
  * Digestive signs: abdominal pain, diarrhoea, constipation, nausea, vomiting
  Edition 2021
  ◌ Cognitive signs using the Q3PC questionnaire (10): memory loss, slowness in reasoning, activity planning or problem solving, concentration, attention difficulties
Other: Outpatient clinic — During a day hospitalization planned during the teleconsultation, patients will benefit from the following multidisciplinary assessment.
  * General clinical examination
  * Assessment of the state of health
  * Respiratory assessment
  * Pulmonary CT assessment
  * Cognitive evaluation
  * Cardiological evaluation
  * Renal assessment
  * Immunological evaluation

SUMMARY:
From July to September 2020, in a first uncontrolled cohort study, 478 patients who were hospitalized at Bicêtre hospital for COVID-19 and who survived were evaluated at 4 months (publication accepted at JAMA). The current project aims to bring together the means to continue this work during the 2nd epidemic wave.

DETAILED DESCRIPTION:
From 15th July to 18th September, 2020, in a first uncontrolled cohort study (Multi-Expertise Consultation of Bicêtre After Covid-19, COMEBAC), we evaluated at four months the surviving patients who were hospitalized at the Bicêtre hospital for COVID-19 during the 1st wave of the epidemic in France and having survived this hospitalization. This cohort included 478 patients. The article resulting from the analysis of the data collected is accepted for publication in JAMA.

This evaluation, the aim of which was both clinical and scientific, was carried out largely thanks to human and material resources then demobilized because of the epidemic and thanks to the investment of doctors and psychologists who carried out the work in addition to their usual work.

The response to the current call for projects aims to bring together the means to continue this monitoring work during the 2nd epidemic wave, while the means and staff are this time completely mobilized by the care of patients with COVID-19 and other. It also aims to raise funds that will allow an in-depth analysis of the residual symptoms presented by the patients.

The current project aims to continue the work started with the COMEBAC "1st wave" cohort with:

* The inclusion of patients hospitalized after the 1st wave.
* An assessment of symptoms according to the SARS-CoV-2 variant.
* A 12-month follow-up of symptomatic patients during the evaluation in COMEBAC "1st wave".

ELIGIBILITY:
For the 6-month evaluation of patients from the 2nd epidemic wave

* Inclusion criteria

  * Age ≥18 years old
  * COVID-19 defined either by a reverse transcriptase-polymerase chain reaction (RT-PCR) or by a combination of clinical signs and compatible lung CT scan
  * Hospitalization for COVID-19 after 1st July 2020
  * Living out of the hospital
* Exclusion criteria

  * Death occurring between index hospitalization and reassessment
  * Patient refusal
  * Discovery of a positive RT-PCR for SARS-CoV-2 during hospitalization for a reason other than COVID-19
  * Nosocomial COVID-19

For the 12-month evaluation of patients from the 1st epidemic wave

* Inclusion criteria

  ◌ Presence of general, cognitive, psychological and respiratory symptoms during the assessment made at 4 months in COMEBAC "1st wave"
* Exclusion criteria

  * Death occurring between the evaluation in COMEBAC "1st wave" and the re-evaluation
  * Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the 1st epidemic wave Patients from the 2nd epidemic wave
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-05-05 (Estimated); Study Completion 2022-05-05 (Estimated)

PRIMARY OUTCOMES:
Prevalence of respiratory, cognitive and psychological symptoms presented at 6 months of hospitalization for COVID-19. | 6 months
  nature and prevalence of symptoms persisting at 6 months of an episode of COVID-19 requiring hospitalization

SECONDARY OUTCOMES:
Difference between the prevalence of residual symptoms between patients hospitalized during the 1st wave of the epidemic in France (from the COMEBAC "1st wave" study) and those of the current study | 6 months
  risk factors for the various sequelae of COVID-19
Association between patient characteristics and the prevalence of residual symptoms. | 6 months
  effect of the therapeutic changes that occurred between the 1st and 2nd wave of COVID-19 on these persistent symptoms.
Association between residual symptoms and the type of SARS-CoV-2 variant | 6 months
  residual symptoms of COVID-19 according to the SARS-CoV-2 variants responsible
Prevalence of respiratory, neurological, cognitive and psychological symptoms presented at 6 months of hospitalization for COVID-19 which occurred during the 1st epidemic wave. | 6 months
  residual symptoms of COVID-19 one year after COVID-19 that occurred during the 1st epidemic wave

CONTACTS AND LOCATIONS:
Overall Officials: Tai PHAM, Principal Investigator — Bicêtre Hospital
Locations (1):
- Bicetre hospital, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No